CLINICAL TRIAL: NCT00243217
Title: Multi-center, Double-blind, Randomized, Placebo-controlled, Six-arm, Parallel-group, Dose-finding Trial to Determine Efficacy, Safety and Tolerability of Five Different Transdermal Doses of Rotigotine in Subjects With Idiopathic Restless Leg Syndrome
Brief Title: Rotigotine Restless Legs Syndrome Dose Finding Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0709
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Idiopathic Restless Leg Syndrome

INTERVENTIONS:
Drug: SPM 936

SUMMARY:
The objective of this trial is to demonstrate clinical efficacy of four different dosages of SPM 962 1.125 mg, 2.25 mg, 4.5 mg and 6.75 mg (corresponding to 2.5 cm2, 5 cm2, 10 cm2 and 15 cm2 patch size respectively) in RLS subjects. It is anticipated that rotigotine (SPM 936) will be more effective than placebo. The tolerability and safety of rotigotine will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Restless Leg Syndrome
* Subject has responded previously, according to medical history information, to L-Dopa therapy and/or treatment with a dopamine agonist, if pre-treated

Exclusion Criteria:

* Secondary restless legs syndrome due to, e.g., renal insufficiency (uremia), iron deficiency anemia, rheumatoid arthritis.
* Secondary restless legs syndrome associated with previous or concomitant therapy with dopamine D2 receptor antagonists, butyrophenones, metoclopramid, atypical antipsychotics (e.g., olanzapine), tri- and tetracyclic antide-pressants, mianserine, lithium or H2-blockers (e.g., cimetidine), or due to withdrawal from drugs such as anticonvulsants, benzodiazepines, barbitur-ates, and other hypnotics.
* History of sleep disturbances like sleep apnea syndrome, narcolepsy, myoclonus epilepsy observed during polysomnography (PSG) or explored in subject history.
* Clinically relevant cardiac dysfunction and/or arrhythmias (e.g., suspected conduction system dysregulations, second or third degree AV block, complete left or right bundle branch block, sick-sinus-syndrome, congestive heart failure Class III or IV by NYHA, myocardial infarction within twelve months prior to enrollment).
* Clinically relevant renal dysfunction (serum creatinine >2.0 mg/dl)
* Clinically relevant hepatic dysfunction (total bilirubin >2.0 mg/dl or ALT and/or AST greater than two times the upper limit of the reference range).
* QTc-interval in resting ECG > 450 msec in males and > 470 msec in females.
* History of symptomatic orthostatic hypotension within 28 days prior to screening visit (Visit 1), or a systolic blood pressure (SBP) less than 105mmHg at trial entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2003-04; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
International RLS Study Group Rating Scale (IRLS): absolute change from baseline to end of maintenance period in the IRLS sum score (difference Visit 7 minus Visit 2)

SECONDARY OUTCOMES:
RLS-6 Rating Scales,CGI (Clinical Global Impressions) - global rating of efficacy by the investigator,Subjective Rating of Efficacy by the subject, Quality of Life. ]

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Schwarz, Monheim, Germany

REFERENCES:
- [Result] Oertel WH, Benes H, Garcia-Borreguero D, Geisler P, Hogl B, Saletu B, Trenkwalder C, Sommerville KW, Schollmayer E, Kohnen R, Stiasny-Kolster K; Rotigotine SP 709 Study Group. Efficacy of rotigotine transdermal system in severe restless legs syndrome: a randomized, double-blind, placebo-controlled, six-week dose-finding trial in Europe. Sleep Med. 2008 Mar;9(3):228-39. doi: 10.1016/j.sleep.2007.04.010. Epub 2007 Jun 5. PMID 17553743